CLINICAL TRIAL: NCT00005977
Title: A Pilot Study of Dose Intensification of Methotrexate in Patients With Advanced-Stage (III/IV) Small Non-Cleaved Cell Non-Hodgkins Lymphoma and B-Cell All
Brief Title: Combination Chemotherapy in Treating Patients With Non-Hodgkin's Lymphoma or Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9917; COG-9917 (Other: Children's Oncology Group); CDR0000067965 (Other: Clinical Trials.gov)
Record Dates: First submitted 2000-07-05; First posted 2003-05-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia; Lymphoma
Keywords: childhood Burkitt lymphoma; L3 childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; Doxorubicin; Etoposide; Ifosfamide; Leucovorin; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- STAGE III NHL (Trt 1) (Experimental): A: Cyclophosphamide (CTX), Doxorubicin hydrochloride, Vincristine sulfate (VCR), Dexamethasone IT Therapy. B: HD-Methotrexate(MTX), Cytarabine(Ara-C), Dexamethasone IT Therapy.
  Treatment ABABA
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: methotrexate; Drug: vincristine sulfate
- STAGE IV NHL, -CNS (Trt 2) (Experimental): A: Cyclophosphamide (CTX), Doxorubicin hydrochloride, Vincristine sulfate (VCR), Dexamethasone IT Therapy. B: HD-Methotrexate(MTX), Cytarabine(Ara-C), Dexamethasone IT Therapy.
  Treatment ABABAB
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: methotrexate; Drug: vincristine sulfate
- STAGE IV, +CNS (Trt 3) (Experimental): A: Cyclophosphamide (CTX), Doxorubicin hydrochloride, Vincristine sulfate (VCR), Dexamethasone IT Therapy. B: HD-Methotrexate(MTX), Cytarabine(Ara-C), Dexamethasone IT Therapy. C: Etoposide, Ifosfamide, Dexamethasone IT Therapy.
  Treatment ABCABAB
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: methotrexate; Drug: vincristine sulfate
- B-ALL, -CNS (Trt 2) (Experimental): A: Cyclophosphamide (CTX), Doxorubicin hydrochloride, Vincristine sulfate (VCR), Dexamethasone IT Therapy. B: HD-Methotrexate(MTX), Cytarabine(Ara-C), Dexamethasone IT Therapy.
  Treatment ABABAB
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: leucovorin calcium; Drug: methotrexate; Drug: vincristine sulfate
- B-ALL, +CNS (Trt 3) (Experimental): A: Cyclophosphamide (CTX), Doxorubicin hydrochloride, Vincristine sulfate (VCR), Dexamethasone IT Therapy. B: HD-Methotrexate(MTX), Cytarabine(Ara-C), Dexamethasone IT Therapy. C: Etoposide, Ifosfamide, Dexamethasone IT Therapy.
  Treatment ABCABAB
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: leucovorin calcium; Drug: methotrexate; Drug: vincristine sulfate

INTERVENTIONS:
Biological: filgrastim — Given IV
  Other Names: GRANULOCYTE COLONY-STIMULATING FACTOR; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
Drug: cyclophosphamide — Given IV
  Other Names: CTX; Cytoxan; NSC #26271; IND #7089
Drug: cytarabine — Given IV
  Other Names: cytosine arabinoside; Ara-C; Cytosar; NSC #638
Drug: dexamethasone — Given IV
  Other Names: DECADRON; NSC #034521
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Adriamycin; NSC #123127; IND #7038
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; NSC #141540; IND #9197
  Arms: B-ALL, +CNS (Trt 3); STAGE IV, +CNS (Trt 3)
Drug: ifosfamide — Given IV
  Other Names: IFX; IFOS; NSC #109724; IND #7887
  Arms: B-ALL, +CNS (Trt 3); STAGE IV, +CNS (Trt 3)
Drug: leucovorin calcium — Given IV
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC #3590
Drug: methotrexate — Given IV
  Other Names: MTX; amethopterin; NSC #740; IND #4291
Drug: vincristine sulfate — Given IV
  Other Names: VCR; Oncovin; NSC #67574; IND #7161

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have non-Hodgkin's lymphoma or acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if increasing the methotrexate dose in combination with standard treatment is feasible in patients with advanced small noncleaved cell non-Hodgkin's lymphoma or B-cell acute lymphocytic leukemia.
* Assess the toxicity of this intensified therapy in these patients.
* Assess the feasibility of treating these patients that have CNS disease at diagnosis with this intensified therapy plus etoposide and ifosfamide.
* Assess toxicities and late effects of this intensive therapy on the central nervous system, cardiac function, and fertility in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to stage and disease (stage III non-Hodgkin's lymphoma (NHL) vs stage IV NHL with no CNS involvement vs stage IV NHL with CNS involvement vs B-cell acute lymphocytic leukemia (B-ALL) with no CNS involvement vs B-ALL with CNS involvement).

Patients receive methotrexate and cytarabine intrathecally on days 1, 4, 11, and 36 (on day 40 for patients with stage IV NHL or B-ALL only) in combination with alternating courses of: A) cyclophosphamide IV every 12 hours for a total of six doses on days 1-3, doxorubicin IV over 30 minutes on day 4, vincristine IV on days 4 and 11, dexamethasone IV or orally twice daily on days 1-5, and filgrastim (G-CSF) subcutaneously (SQ) or IV over 30 minutes beginning on day 5 and continuing until blood counts recover and B) methotrexate IV over 24 hours on day 18, methotrexate intrathecally on day 18, dexamethasone IV or orally twice daily on days 18-22, leucovorin calcium IV or orally every 6 hours for a total of 6 doses on days 20-21, cytarabine IV over 48 hours on days 20-21, and G-CSF SQ or IV over 30 minutes beginning on day 22 and continuing until blood counts recover. Patients with stage III NHL receive at total of 5 courses of treatment (A-B-A-B-A) and patients with stage IV NHL or B-ALL with no CNS involvement receive a total of 6 courses of treatment (A-B-A-B-A-B).

Patients with CNS involvement receive a third course of treatment: C) etoposide IV over 1 hour on days 36-40, ifosfamide IV over 1 hour on days 36-40, oral dexamethasone twice daily on days 36-40, and G-CSF SQ or IV over 30 minutes beginning on day 41 and continuing until blood counts recover. Patients with CNS involvement receive a total of 7 courses of treatment (A-B-C-A-B-A-B).

Patients are followed every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 27-80 patients will be accrued for this study over 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically confirmed small noncleaved cell non-Hodgkin's lymphoma

    * Stage III or IV
    * Burkitt's or non-Burkitt's by the Working Formulation OR
    * Burkitt's or Burkitt's-like by the REAL classification
  * Histologically confirmed B-cell acute lymphocytic leukemia

    * At least 25% blasts in bone marrow
    * FAB L3 morphology
    * FAB L1 morphology allowed if blasts show B-cell markers (CD19, 20, 22) and surface immunoglobulin positivity
    * Must be registered on POG-9900 in past 8 days

PATIENT CHARACTERISTICS:

Age:

* Under 22 at time of diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test
* HIV positive allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent use of dexamethasone as antiemetic

Radiotherapy:

* Not specified

Surgery:

* Prior surgery allowed

Other:

* No prior therapy except surgery

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2000-09; Primary Completion 2004-03 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 1 year
  Assess the effect of high dose methotrexate in combination with standard treatment per the POG 9317 protocol on 1-year event-free survival (EFS), monitor and assess toxicity, and estimate the hospitalization costs for the treatment of toxicity related side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Hazem H. Mahmoud, MD, Study Chair — Carol G. Simon Cancer Center at Morristown Memorial Hospital
Locations (119):
- United States (104):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Children's Hospital and Health Center, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - University of Miami-Jackson Memorial Hospital Medical Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Texas Oncology P.A., Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School-Charleston, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Royal Children's Hospital, Parkville, Victoria, Australia
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Laval University Medical Center, Sainte-Foy, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Clinique de Pediatrie, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne